CLINICAL TRIAL: NCT00228605
Title: An Open-Label 12 Month Study to Evaluate the Safety, Tolerability and Efficacy of OraVescent Fentanyl Citrate for the Management of Breakthrough Pain in Opioid-Tolerant Patients With Chronic Noncancer Pain
Brief Title: Evaluating the Safety and Tolerability of OraVescent Fentanyl for Opioid Tolerant Patients With Noncancer Related Breakthrough Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cephalon (Industry)
Organization: Teva Branded Pharmaceutical Products R&D, Inc. (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C25608/3040/BP/US
Record Dates: First submitted 2005-09-27; First posted 2005-09-29 (Estimated); Last update posted 2014-05-09 (Estimated); Status verified 2014-05

CONDITIONS: Low Back Pain; Migraine; Diabetic Neuropathies; Osteoarthritis
Keywords: Pain; Sudden Pain; Flares; noncancer; low back pain; neuropathic pain; osteoarthritis pain; migraine; chronic headache; diabetic peripheral neuropathy
MeSH Terms: conditions — Low Back Pain; Migraine Disorders; Diabetic Neuropathies; Osteoarthritis; Pain; Neuralgia; Headache Disorders

INTERVENTIONS:
Drug: OraVescent Fentanyl

SUMMARY:
The purpose of this study is to evaluate the safety and tolerability of OraVescent fentanyl for the potential treatment of breakthrough pain episodes in patients who have chronic noncancer pain.

ELIGIBILITY:
Inclusion Criteria:

* Chronic pain diagnosis
* Opioid tolerant
* Has on average 1-4 breakthrough pain episodes per day

Exclusion Criteria:

* Drug abuse history
* Cardiopulmonary disease
* Monoamine oxidase inhibitors (MAOIs)
* Expected to have surgery to relieve the pain

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500
Dates: Start 2005-03; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Safety and tolerability when used over a 12-month period for the management of breakthrough pain in opioid tolerant patients

SECONDARY OUTCOMES:
Assess the patients' quality of life through questionnaires
Assess the patients' overall medication preferences
Assess the patients' overall medication performance

CONTACTS AND LOCATIONS:
Overall Officials: Gwendolyn Neibler, DO, Study Director — Cephalon
Locations (38):
- United States (38):
  - MedSearch, Calera, Alabama
  - Clinical Research Consultants, Inc., Hoover, Alabama
  - Arizona Research Center, Phoenix, Arizona
  - NEA Clinic, Jonesboro, Arkansas
  - Lynn Institute of the Rockies, Colorado Springs, Colorado
  - Radiant Research-Daytona Beach, Daytona Beach, Florida
  - Advent Clinical Research Centers, Inc., St. Petersburg, Florida
  - Gold Coast Research, Weston, Florida
  - Center for Prospective Outcome Studies, Inc., Atlanta, Georgia
  - Advent Clinical Research Centers, Inc., Atlanta, Georgia
  - Center for Prospective Outcome Studies, Inc., Marietta, Georgia
  - North Fulton Regional Hospital Pain Center, Roswell, Georgia
  - Carmen Research, Smyrna, Georgia
  - Orthopedic Health Care, Boise, Idaho
  - Medisphere Medical Research Center, LLC, Evansville, Indiana
  - Tri-State Arthritis & Rheumatology Center, LLC, Evansville, Indiana
  - Iowa Pain Management Clinic, PC, Des Moines, Iowa
  - Mid-America Physiatrists, PA, Overland Park, Kansas
  - Capital Clinical Research Associates, LLC, Rockville, Maryland
  - Brigham Women's Hospital, Attn: Pain Trials Center, Boston, Massachusetts
  - MedVadis Research, Wellesley Hills, Massachusetts
  - Medex Healthcare Research Center, St Louis, Missouri
  - Radiant Research - St. Louis, St Louis, Missouri
  - Clinical Research Center of Nevada, Las Vegas, Nevada
  - Northshore University Hospital, Bethpage, New York
  - NYU Pain Management Center, New York, New York
  - Research Across America, New York, New York
  - The Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Southern Oregon Health & Wellness, Medford, Oregon
  - Clinical Research Center of Reading, LLP, West Reading, Pennsylvania
  - Healthstar Physicians, Morristown, Tennessee
  - Biopharma Research Associates, Sugar Land, Texas
  - Lifetree Clinical Research, Salt Lake City, Utah
  - Radiant Research, Salt Lake City, Utah
  - Huntsman Cancer Institute, Salt Lake City, Utah
  - Pain Management Center, South Burlington, Vermont
  - Northwest Clinical Research Center, Bellevue, Washington
  - Rowan Research, Spokane, Washington